CLINICAL TRIAL: NCT02579005
Title: Radio-Immuno-Modulation for Advanced Lung Cancer: a Pilot Study Evaluating Tolerance and Immune Responses
Brief Title: Radio-Immuno-Modulation in Lung Cancer
Acronym: RIM
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of ressources
Sponsor: Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal (Other)
Collaborators: Maisonneuve-Rosemont Hospital (Other)
Responsible Party: Principal Investigator, Dr. Razvan Bucur Diaconescu, Hematologist-Oncologist, Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-634
Record Dates: First submitted 2015-10-07; First posted 2015-10-19 (Estimated); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Lung Cancer
Keywords: Radiation; Immune response; Anti-tumor; Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients with a living donor (Experimental): Radiation + PBMC
  Interventions: Biological: Patients with a living donor
- Patients with a UCB donor (Experimental): Radiation + UCB
  Interventions: Biological: Patients with a UCB donor

INTERVENTIONS:
Biological: Patients with a living donor — The day of allogeneic cell infusion will be referred to as Day 0 and the n-th day before that, as Day -n. The dose of external radiation will be 15 Gy divided in 3 fractions, from Day -3. Cyclophosphamide, 250 mg/m2 will be given on Day -2. Donors will receive 5 daily doses of GCSF, 10 µg/kg, by subcutaneous injection from Day -4. PBMC will be collected through apheresis on Day 0. A dose of 5 x 10exp7 CD3 cells/kg will be administered. The infused volume will be adjusted to contain this T cell dose.
  Arms: Patients with a living donor
Biological: Patients with a UCB donor — The day of allogeneic cell infusion will be referred to as Day 0 and the n-th day before that, as Day -n. The UCB unit should have at least 4 of 6 HLA compatibility and at least 3 x 10exp6 TNC per kg patient weight. The dose of external radiation will be 15 Gy, divided in 3 fractions, starting on Day -3. Cyclophosphamide, 250 mg/m2 intravenously, will be given on Day -2.
  Arms: Patients with a UCB donor

SUMMARY:
This project will assess the feasibility of treating advanced cancer using the immune system, without any anti-cancer drug. In this pilot study, the investigators propose combining low-dose radiotherapy, in lung cancer patients, with allogeneic immune cells obtained from a donor. The patients will receive radiotherapy directed to one of the patient's tumors, as well as an immunomodulatory drug called cyclophosphamide. Thereafter, they will receive the infusion of donor immune cells.

DETAILED DESCRIPTION:
Metastatic lung cancer remains incurable despite numerous studies and treatments tried, including chemotherapy and, more recently, targeted therapies.

Cancer can escape immune surveillance through different mechanisms: low levels of tumor associated antigens (TAA), regulatory T cells, and immunosuppressive cytokines. Non-cytolytic doses of radiation have been shown to reverse some of these pathways in experimental models. It up-regulated the density of the MHC molecules presenting TAA and increased the T cell infiltration of the tumor (1). Patients with lymphoma, liver or prostate cancer were treated with radiotherapy combined with immunotherapy, in the form of a TLR9 agonist, autologous dendritic cells or a prostate-specific antigen vaccine (2, 3, 4). These trials have shown an induction of T cell reactivity against TAA. Another form of immunotherapy, used for patients with refractory hematologic malignancies is allogeneic hematopoietic stem cell transplantation (HSCT) (5). Its success has relied on cell infusions from a donor, demonstrating the immunologic control sustained by allogeneic cells (6).

The approach investigated in this study uses the immune cells from a donor to induce a tumor destruction reaction. This will be amplified by the immunological effects of radiotherapy. Many oncogenes are present in lung cancers and low-dose radiation increases their expression on the surface of the tumor cell. In addition, radiation has the property to stimulate the production of inflammatory cytokines and chemokines in the irradiated site. Finally, the donor's immune cells shall respond physiologically by migrating to the site of inflammation. This will trigger an immune reaction directed against the abnormal cancer cells.

A total of 24 patients are expected to be recruited over the study period, estimated to be 3 years. The allogeneic cells will be obtained from one of two possible donor types. For patients having a living donor, the immune cells will be harvested through a collection procedure called apheresis. The living donor should be a sibling with 3/6 or less HLA compatibility with the patient, at the A, B and DRB1 loci. For patients who do not have such a living donor, allogeneic cells from a cryopreserved umbilical cord blood (UCB) unit will be used.

The treatment course will be the following: low-dose radiotherapy will be delivered to a single tumor site, which could be either the primary tumor or one of its metastases. Low-dose cyclophosphamide will be given to decrease regulatory T cell activity and increase anti-tumor responses. Allogeneic immune cells will be administered thereafter, according to the treatment arm the patient has been assigned.

ELIGIBILITY:
Inclusion criteria:

* Advanced lung cancer documented by a histo-pathological analysis;
* Patients who received at least one line of anti neoplastic therapy;
* Presence of at least one tumor mass >1 cm and not previously irradiated;
* Metastases situated in one of the following sites: lung, skeleton, lymph nodes or soft tissue;
* Presence of at least one not previously irradiated metastasis;
* Life expectancy greater than 3 months;
* ECOG performance status ≤ 2.

Exclusion criteria:

* Second active cancer necessitating treatment;
* History of autoimmune disease;
* Patients dependent on immunosuppressive medications, including corticosteroids;
* Decreased diffusion capacity below 40%, if radiation planned to a lung metastasis;
* Patients needing urgent radiotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2018-04-20 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-related adverse events | Up to 6 months
  Evaluation by follow-up clinic visits, including medical questionnaire, physical exam & blood tests: complete blood count, electrolytes, renal & liver function tests. AE will be graded using National Cancer Institute's Common Toxicity Criteria version 3 (7). Evaluations will take place twice a week for the first 2 weeks, weekly for 2 weeks, every 2 weeks for 2 months & every month for 3 months. It is anticipated that a maximum of 1 of 6 patients will have grade 3 side effects, including nausea, diarrhea, dyspnea, cough, fever, rash.

SECONDARY OUTCOMES:
Immune responses - T cell infiltration | Up to 1 month
  Assessment using biopsies done before & 1-2 weeks after treatment. The block slides will be stained with CD3, CD4, CD8 & PDL-1 antibodies. T cell density will be expressed as the number of CD4+ and CD8+ cells to tumor cell ratio. The degree of T cell infiltration of the tumors will be assessed by comparing these ratios between pre & post treatment samples.
Immune responses - Tumor cell phenotype | Up to 1 month
  Assessment using biopsies done before & 1-2 weeks after treatment. Flow cytometry will be used to assess the following tumor markers: HLA, Fas, ICAM-1, PDL-1. The changes in tumor cell phenotypes will be assessed by comparing the mean fluorescence intensity of the above markers between pre & post treatment samples. The PDL-1 tumor cell expression will also be compared on the block slides between pre & post treatment samples.
Immune responses - tumor infiltrating T cell phenotype | Up to 1 month
  Assessment using biopsies done before & 1-2 weeks after treatment. Flow cytometry will be used to assess the following markers on tumor infiltrating T cells: CD3, CD4, CD8, CD25 & Foxp3. The nature and magnitude of T cell infiltration will be assessed by comparing the frequencies of these T cell subsets between pre & post treatment samples.
Immune responses - origin of tumor infiltrating T cells | Up to 1 month
  Assessment using biopsies done 1-2 weeks after treatment. Single cell suspensions will be stained with the following markers for tumor infiltrating T cells: CD3, CD4 and CD8. CD4+ and CD8+ T cells will be isolated by fluorescence-activated cell sorting. Their origin (patient vs donor) will be determined by a chimerism assay. The frequencies of donor-derived cells will be determined by PCR quantification of patient and donor specific VNTR bands.

CONTACTS AND LOCATIONS:
Overall Officials: Razvan B Diaconescu, MD, Principal Investigator — CIUSSS du Nord-de-l'Île-de-Montréal - Hôpital du Sacré-Cœur de Montréal
Locations (1):
- Hopital Sacre-Coeur, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hodge JW, Guha C, Neefjes J, Gulley JL. Synergizing radiation therapy and immunotherapy for curing incurable cancers. Opportunities and challenges. Oncology (Williston Park). 2008 Aug;22(9):1064-70; discussion 1075, 1080-1, 1084. PMID 18777956
- [Background] Brody JD, Ai WZ, Czerwinski DK, Torchia JA, Levy M, Advani RH, Kim YH, Hoppe RT, Knox SJ, Shin LK, Wapnir I, Tibshirani RJ, Levy R. In situ vaccination with a TLR9 agonist induces systemic lymphoma regression: a phase I/II study. J Clin Oncol. 2010 Oct 1;28(28):4324-32. doi: 10.1200/JCO.2010.28.9793. Epub 2010 Aug 9. PMID 20697067
- [Background] Chi KH, Liu SJ, Li CP, Kuo HP, Wang YS, Chao Y, Hsieh SL. Combination of conformal radiotherapy and intratumoral injection of adoptive dendritic cell immunotherapy in refractory hepatoma. J Immunother. 2005 Mar-Apr;28(2):129-35. doi: 10.1097/01.cji.0000154248.74383.5e. PMID 15725956
- [Background] Gulley JL, Arlen PM, Bastian A, Morin S, Marte J, Beetham P, Tsang KY, Yokokawa J, Hodge JW, Menard C, Camphausen K, Coleman CN, Sullivan F, Steinberg SM, Schlom J, Dahut W. Combining a recombinant cancer vaccine with standard definitive radiotherapy in patients with localized prostate cancer. Clin Cancer Res. 2005 May 1;11(9):3353-62. doi: 10.1158/1078-0432.CCR-04-2062. PMID 15867235
- [Background] Diaconescu R, Storb R. Allogeneic hematopoietic cell transplantation: from experimental biology to clinical care. J Cancer Res Clin Oncol. 2005 Jan;131(1):1-13. doi: 10.1007/s00432-004-0611-6. Epub 2004 Sep 28. PMID 15565456
- [Background] Baron F, Maris MB, Sandmaier BM, Storer BE, Sorror M, Diaconescu R, Woolfrey AE, Chauncey TR, Flowers ME, Mielcarek M, Maloney DG, Storb R. Graft-versus-tumor effects after allogeneic hematopoietic cell transplantation with nonmyeloablative conditioning. J Clin Oncol. 2005 Mar 20;23(9):1993-2003. doi: 10.1200/JCO.2005.08.136. PMID 15774790
- [Background] 7. Cancer Therapy Evaluation Program. Common Terminology Criteria for Adverse Events v3.0 (CTCAE). Bethesda, MD. National Cancer Insitute, 2006. Available at: http://ctep.cancer.gov/protocolDevelopment/electronic_applications/docs/ctcaev3.pdf.